CLINICAL TRIAL: NCT00380211
Title: A Randomized, Double-Blind Trial Evaluating the Safety and Immunogenicity of an Influenza Vaccine With Reduced Preservative (FluLaval™ TR) and a Standard Influenza Vaccine (Fluarix®) in Subjects Between 18-60 and Over 60 Years of Age.
Brief Title: Safety and Immunogenicity of FluLaval™ TR and Fluarix® (Influenza Vaccines) in Young and Older Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IDB-200-001
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Influenza
Keywords: Thimerosal reduced content; Immunogenicity, safety, reactogenicity; Young and elderly adults; Influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; fluarix

INTERVENTIONS:
Biological: Influenza vaccine (A/H3N2, A/H1N1, and B strains)
Biological: Fluarix

SUMMARY:
The purpose of this trial is to describe the immunogenicity, the safety, and tolerability of FluLaval™ TR and Fluarix®, the latter serving as active comparator. The results will be compared to a standard immune response criteria, for both young and elderly populations.

DETAILED DESCRIPTION:
This randomized trial will assess the immune protection offered at Day 21 by FluLaval™ TR, Fluarix® being the comparator. In both groups, immune response will be assessed through a blood test before and 21 days following vaccination. The safety and tolerability of the study vaccine will be contrasted to the comparator vaccine over a period of 42 days following vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults (≥18 yrs)
* Stable health status
* Provide informed consent
* Access to direct phone service (NOT a pay phone or a common-use phone service)
* Eligible females must have a negative pregnancy test

Exclusion Criteria:

* Febrile illness (>38.0°C oral temperature)
* High blood pressure (≥140/90 mmHg)
* Significant acute or chronic
* Uncontrolled medical or psychiatric illness within 1 month prior to vaccination
* Immunosuppressive condition (confirmed or suspected)
* Renal impairment
* Hepatic dysfunction
* Complicated insulin-dependent diabetes mellitus
* Unstable cardiopulmonary disease
* Blood dyscrasias
* Cytotoxic, immunosuppressive drug, or glucocorticoids use within 1 month of vaccination (nasal glucocorticoids allowed)
* History of demyelinating disease
* Active neurological disorder
* Significant alcohol or drug abuse
* Significant coagulation disorder (prophylactic antiplatelet medications allowed)
* Influenza vaccine administrated within 6 months prior to study vaccination
* Administration of any other vaccine from 30 days prior to the end of the study
* Use of non-registered drug within 30 days prior to study vaccination
* Receipt of immunoglobulins and/or any blood products within 3 months of study vaccination
* History or suspected allergy to previous influenza vaccine, or to any constituent of FluLaval™ TR and Fluarix®, or reaction to eggs consumption
* Pregnant or nursing female subjects
* Female subjects not protected by an acceptable contraception method (except if surgically sterile or post-menopausal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2006-09; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
21 days after vaccination: seroconversion rate, seroprotection rate,
geometric mean titer fold increase

SECONDARY OUTCOMES:
Immediate AEs; solicited and spontaneous AEs within 42 days of vaccination;
SAEs over the whole study period

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- United States (6):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Binghamton, New York
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Burke, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: IDB-200-001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: IDB-200-001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: IDB-200-001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: IDB-200-001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: IDB-200-001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register